CLINICAL TRIAL: NCT01282216
Title: Patient-donor Vaccination in the Context of Allogeneic Bone Marrow Transplant (BMT) With High-dose Post Transplantation Cyclophosphamide.
Brief Title: Patient-donor Vaccination in the Context of Allogeneic Bone Marrow Transplant With Post-transplant Cyclophosphamide
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual and loss of funding.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: J10140; P01CA015396 (NIH); NA_00044665 (Other: JHM IRB)
Record Dates: First submitted 2011-01-13; First posted 2011-01-24 (Estimated); Results first posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Transplant-Related Cancer
MeSH Terms: interventions — Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Only the study pharmacist was unblinded.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Donor PCV13 (Active Comparator): Donors receive PCV13 prior to bone marrow donation.
  Interventions: Biological: PCV13
- Donor Havrix (Active Comparator): Donors receive Havrix prior to bone marrow donation.
  Interventions: Biological: Havrix
- Recipient vaccine (Active Comparator): Recipients receive Havrix and PCV13 post bone marrow transplant.
  Interventions: Biological: Havrix; Biological: PCV13

INTERVENTIONS:
Biological: Havrix — 1440 ELISA units, or 1 mL, IM
  Other Names: Hepatitis A vaccine
  Arms: Donor Havrix; Recipient vaccine
Biological: PCV13 — 0.5 mL IM
  Other Names: Prevnar-13
  Arms: Donor PCV13; Recipient vaccine

SUMMARY:
This research is being done to understand the effects of certain types of bone marrow transplant (BMT) on the immune system. Your doctors are planning a BMT, using one of your family members as the bone marrow donor, for your cancer. Part of that BMT involves a chemotherapy drug, called Cyclophosphamide (Cytoxan), given after the transplant. This research is being done to understand the effects of Cyclophosphamide on the immune system.

DETAILED DESCRIPTION:
The research will involve giving your donor a vaccine against a certain infection, before the bone marrow donation: either a vaccine against hepatitis (the hepatitis A vaccine), or a vaccine against pneumonia (Prevnar). You will then get both of these vaccines following your transplant. By studying how much these vaccines may improve your immune system, we hope to better understand the effects of the BMT with Cyclophosphamide on the immune cells.

Prevnar is a pneumococcal vaccine (pneumococcus is a bacteria that can cause pneumonia and other infections). It is approved by the Food and Drug Administration (FDA) for the prevention of infections in children. It is not usually given to adults. Hepatitis A vaccine is approved by the FDA for the prevention of hepatitis A (a liver infection) in children and adults.

The vaccines are not approved for bone marrow donors or for vaccinating adults after BMT (using these vaccines in this research is investigational). The FDA is allowing the use of these vaccines in this research study.

Certain people getting BMT followed by Cyclophosphamide may join, if their donors might also join. Your bone marrow donor must take part in this study, in order for you to continue on this study

ELIGIBILITY:
Inclusion Criteria:

Patients inclusion for study:

1. Patient age > 18 years.
2. Plan to undergo one of the following types of transplant, using bone marrow from a related donor:

   * Myeloablative, HLA matched or partially HLA-mismatched (haploidentical), related-donor bone marrow transplantation that includes high-dose posttransplantation Cy
   * Nonmyeloablative, HLA matched or partially HLA-mismatched, related-donor bone marrow transplantation that includes high-dose posttransplantation Cy Note: Patients who receive posttransplantation rituximab are eligible.

Patients inclusion for vaccine:

1. Receipt of the type of myeloablative or nonmyeloablative BMT
2. The bone marrow donor has received the pre-bone marrow harvest vaccine (either Prevnar or hepatitis A vaccine) on this study.

Donors inclusion:

1. Donor age > 18 years.

Exclusion Criteria:

Patients exclusion for study entry:

1. Hypersensitivity to either the components of hepatitis A vaccine (including neomycin) or the components of the PCV7 and PCV13 vaccines (including diphtheria toxin).
2. Severe latex allergy.

Patients exclusion for vaccine:

1. Graft failure.
2. Disease progression or relapse, or disease persistence requiring treatment.Note: Patients with asymptomatic or low-volume disease progression or relapse may be eligible, determined on a case-by-case basis by the PI.
3. Systemic immunosuppression for GVHD treatment or prophylaxis within 4 weeks (+/- 5 days) prior to vaccination.
4. Pregnant or breastfeeding

Donors exclusion:

1. Hypersensitivity to both the components of hepatitis A vaccine (including neomycin) and the components of the PCV7 and PCV13 vaccines (including diphtheria toxin).
2. Severe latex allergy.
3. Expected to be on systemic immunosuppressants between the time of vaccination and the bone marrow donation.
4. Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: RIchard Ambinder, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8 recipients and 8 donors were screen failures prior to starting the study. 8 additional donors were vaccinated, but their intended recipients were never vaccinated and were replaced on study due to early relapse or graft failure. Data for the latter 8 donors has been lost and their arm assignment cannot be determined.
Groups:
- Donor - Assignment Unknown: Donors in this group received either PCV13 or Havrix. Assignment cannot be determined due to missing study data.
Period: Overall Study
Arm/Group | Donor PCV13 | Donor Havrix | Recipient Vaccine | Donor - Assignment Unknown
Started | 18 | 26 | 52 | 8
Completed | 18 | 26 | 19 | 0
Not Completed | 0 | 0 | 33 | 8
Not completed — Graft failure | 0 | 0 | 3 | 2
Not completed — Physician Decision | 0 | 0 | 11 | 0
Not completed — Relapse | 0 | 0 | 17 | 6
Not completed — Death | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Data for 8 donors has been lost and their arm assignment cannot be determined; therefore, donor vaccine arms/groups are combined in this module.
Groups:
- Donor Vaccine: Donors are randomized to receive either Havrix or PCV13 prior to bone marrow donation.
- Total: Total of all reporting groups
Arm/Group | Donor Vaccine | Recipient Vaccine | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 44 | 94
  >=65 years | 2 | 8 | 10
Age, Continuous [Median (Full Range); unit: years] | 41.5 [19 to 72] | 54 [19 to 70] | 50 [19 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 31 | 30 | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 52 | 104

OUTCOME MEASURES:

1. Primary Outcome: T-cell Immunity Augmentation
Description: Number of participants in which patient-donor pairs were not pre-immune to hepatitis A or CRM197, show augmented T-cell immunity when the vaccine is also given to the bone marrow donor.
Time Frame: up to 6 months
Population: Samples collected were inadequate for analysis, therefore data could not be collected to assess this outcome measure.
Arm/Group | Donor Vaccine | Recipient Vaccine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Recipient Vaccine-specific T-cell Response Post-transplant, Before Vaccination
Description: Number of participants with a greater T-cell response after receiving transplant from a donor who received a vaccine, before receiving post-transplant vaccination.
Time Frame: up to 6 months
Population: Samples collected were inadequate for analysis, therefore data could not be collected to assess this outcome measure.
Arm/Group | Donor Vaccine | Recipient Vaccine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Recipient Vaccine-specific T-cell Response After Post-transplantation Vaccine
Description: Number of participants with a greater T-cell response after receiving transplant from a donor who received a vaccine, and after receiving post-transplant vaccination.
Time Frame: up to 6 months
Population: Samples collected were inadequate for analysis, therefore data could not be collected to assess this outcome measure.
Arm/Group | Donor Vaccine | Recipient Vaccine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 1 month
Description: Only unexpected or serious adverse events that were considered related to either vaccine were tracked and reported. Adverse events were captured systematically by investigator assessment for at least 10 days for donors and at least 28 days for recipients. Data for 8 donors has been lost and their arm assignment cannot be determined, therefore donor vaccine arms/groups are combined in this module
Arm/Group | Donor Vaccine | Recipient Vaccine
All-Cause Mortality (participants affected / at risk) | 0/52 | 2/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes